CLINICAL TRIAL: NCT04135508
Title: A Multicenter, Randomized, Double-Blind, Phase III Clinical Trial Parallel Controlled With Humira to Evaluate the Efficacy and Safety of BAT1406 Injection in the Treatment of Ankylosing Spondylitis
Brief Title: A Phase III Study Evaluate the Efficacy and Safety of BAT1406 and Humira
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-1406-003-CR
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAT1406 (Experimental): Adalimumab, 40 mg/0.8 mL/vial, subcutaneously 1 vial every two weeks, up to a maximum of 6 months treatment.
  Interventions: Drug: BAT1406
- Humira (Active Comparator): Adalimumab, 40 mg/0.8 mL/vial, subcutaneously 1 vial every two weeks, up to a maximum of 6 months treatment.
  Interventions: Drug: Humira

INTERVENTIONS:
Drug: BAT1406 — 40mg/0.8ml
  Other Names: No Other Intervention Names
  Arms: BAT1406
Drug: Humira — 40mg/0.8ml
  Other Names: Adalimumab
  Arms: Humira

SUMMARY:
A Phase III Study Evaluate the Efficacy and Safety of BAT1406 and Humira

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, active comparator, parallel two arm study to compare the efficacy, and to evaluate the safety, and immunogenicity of BAT1406 to Humira® in patients with active ankylosing spondylitis (AS) to demonstrate clinical equivalence of BAT1406 and Humira®.

ELIGIBILITY:
Inclale or female. usion Criteria: 1.Must be between 16-65 years old (inclusive) at the time of signing the ICF; 2.Subjects must meet the diagnostic criteria for AS (AS New York standard revised in 1984) by providing pelvic X-rays taken within six months prior to enrollment.

3.Subjects suffer from active AS during screening. Active AS is defined as: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) ≥ 4, spinal pain ≥ 4.

4.Subjects' liver and kidney function indicators should meet the following requirements during screening:

a. Serum creatinine (Cr) < 1.7 × upper limit of normal (ULN), or creatinine clearance (CCr) > 75 mL/min.

b.Alanine Transaminase (ALT) < 2 × ULN. c.Aspartate Transaminase (AST) < 2 × ULN. 5.The subjects' hematology laboratory test indicators meet the following requirements during screening:

1. Hemoglobin ≥ 8.0 g/dL.
2. White blood cell count ≥ 3.5 × 109/L.
3. Neutrophil count ≥ 1.5×109/L.
4. Platelet count ≥ 100×109/L. 6.Prior to screening, subjects were allowed to use stable doses of MTX (≤ 25 mg/week), sulfasalazine (< 3 g/day), NSAIDs, and/or analgesics, but the doses should have been stabled for at least 4 weeks prior to screening, and must remain unchanged during the trial.

   7.Prior to screening, subjects were allowed to use glucocorticoids, but are limited to daily oral doses of prednisone of ≤ 10 mg or equivalent. Doses should have been stable for at least 4 weeks prior to screening, and should remain unchanged during the trial. In addition, subjects were permitted to use topical/ophthalmic/otic medications containing low potency glucocorticoids according to product monographs.

   8.Subjects discontinuing leflunomide should have been treated with cholestyramine (8 grams each time, t.i.d) for 11 days, and there should have been a 4-week washout period from the first dose of cholestyramine. For subjects discontinuing leflunomide and not treated with cholestyramine, a 12-week washout period from the last dose of leflunomide to the screening period was required.

   9.During screening, if the subjects were using botanical preparations (such as Tripterygium Wilfordii, total glucosides of paeony, sinomenine, yishen juanbi pill, etc.) for the treatment of AS, or thalidomide, or were treated with physical therapy, they should have stopped these medications and treatments for at least 4 weeks before being considered eligible candidates.

   10.During screening, if the subjects had previously received live (attenuated) virus/bacterial vaccines, or had received intravenous injection of immunoglobulin IgG, they must have stopped the medications for at least 12 weeks before being considered eligible for enrollment.

   11.Women of childbearing age must have had a negative serum and/or urine pregnancy test prior to enrollment, and must not have been breastfeeding.

   12.Subjects of childbearing age (regardless of gender) must have voluntarily agreed to use reliable contraceptive methods (except for non-fertile women and men who have undergone vasectomy) from signing of the ICF to 6 months after the last dose of treatment. Contraceptive methods include but are not limited to: hormonal contraception, physical contraception, or abstinence.

Note: During screening, women who have entered menopause for less than 12 continuous months or men who have undergone vasectomy within 6 months should use reliable contraception methods.

13.Subjects should have the ability to understand the nature and purpose of the trial, including possible risks and side effects, be able to understand the verbal and written instructions given by the investigators, and can follow the requirements of the trial.

14.Subjects voluntarily sign the ICF.

Exclusion Criteria:

1. Subjects have used any biological products to treat AS within 6 months prior to the enrollment.
2. Clinical or imaging studies suggested that the spine has reached complete rigidity (if there were two consecutive lumbar vertebrae not fused together, then the spine has not reached complete rigidity).
3. Allergic to any ingredients of Humira, allergic to human proteins or susceptible to immunoglobulin allergies.
4. Subjects with a medical history of hepatitis B, hepatitis C, HIV, any immunodeficiency, or with a positive laboratory test result (hepatitis B surface antigen, hepatitis C antibody, or HIV antibody) during screening.
5. Subjects diagnosed with active pulmonary tuberculosis, latent tuberculosis infection, or subjects suspected of tuberculosis based on clinical manifestations (including but not limited to pulmonary tuberculosis).
6. Subjects with positive T.SPOT.TB test or abnormalities in tuberculosis-related chest X-ray; or subjects with TB who have not received standard treatment of at least 30 days.
7. Active infections, including acute and chronic infections, and local infections (such as sepsis, abscesses, opportunistic infections, and invasive fungal infections).
8. Subjects who have taken oral antibiotics within 2 weeks prior to the screening or have been given intramuscular/intravenous treatments for infection within 4 weeks prior to the screening, or have had severe infections within 6 months prior to the screening (investigators must determine the potential risks of subjects' enrollment based on the individual's clinical history).
9. Subjects with a history of recurrent herpes zoster, history of Listeria infection, reticuloendotheliosis, and other chronic or recurrent infections.
10. Subjects who have undergone ostectomy/arthrectomy/synovectomy within 3 months prior to the screening, or planned to undergo joint or spinal surgery during the trial.
11. Subjects with clinically significant laboratory abnormalities that suggested the presence of unknown disease and required further clinical examination.
12. Subjects with an apparent history of drug abuse or alcohol dependence at present or in the past 2 years.
13. Subjects with one or more of the following diseases:

    1. Subjects without self-care ability, those who require wheelchairs or those who are bedridden;
    2. Uncontrolled hypertension (defined as systolic pressure >150 mmHg, or diastolic pressure >100 mmHg during the screening period);
    3. Subjects with a history of congestive heart failure (New York Heart Association classification III/IV);
    4. Subjects with a history of acute myocardial infarction or unstable angina within 12 months prior to the screening;
    5. Subjects with serious arrhythmias;
    6. Any subject with clinically significant respiratory diseases, including but not limited to chronic obstructive pulmonary disease, asthma, interstitial lung disease, bronchiectasis, and pleural effusion;
    7. Subjects with a history of demyelinating diseases or with symptoms suggestive of such diseases, including but not limited to: multiple sclerosis and Guillain-Barré syndrome;
    8. Subjects who had not used a stable dose of medication to control diabetes within 4 weeks prior to the screening (glycated hemoglobin HbA1c >7% during screening);

    h.Subjects with any arthritis or rheumatic diseases (in addition to AS) that may affect the evaluation of the clinical study, including but not limited to: rheumatoid arthritis, osteoarthritis, psoriatic arthritis, systemic lupus erythematosus, gouty arthritis, and fibromyalgia; j.Subjects with any neurological, psychotic, or other systemic diseases that may affect the clinical efficacy evaluation; k.Subjects who have had a history of malignancy in the past 5 years (except for non-metastatic squamous cell carcinoma or basal cell carcinoma or cervical carcinoma in situ that have been cured); l.History of lymphoma or lymphoproliferative diseases.
14. Subjects using the following concomitant drugs:

    1. Have used alkylating preparations within 12 months prior to the screening.
    2. Injected corticosteroids into the joint cavity, muscle or vein within 4 weeks prior to screening.
15. Subjects who have participated in other clinical trials within 3 months prior to the enrollment or planned to participate in other clinical trials.
16. The investigator determined that the subject was not suitable for this trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment in SpondyloArthritis international Society (ASAS) 20 | week 12
  the percentage of subjects achieving the Assessment in SpondyloArthritis international Society (ASAS) 20 treatment response

SECONDARY OUTCOMES:
Percentage of subjects achieving ASAS20 treatment response | week 24
  the percentage of subjects achieving the Assessment in SpondyloArthritis international Society (ASAS) 20 treatment response
Percentage of subjects achieving ASAS40 treatment response | week 12; week 24
  the percentage of subjects achieving the Assessment in SpondyloArthritis international Society (ASAS) 40 treatment response
Percentage of subjects achieving ASAS5/6 treatment response | week 12; week 24
  the percentage of subjects achieving ASAS5/6 treatment response
Percentage of subjects achieving BASDAI50 treatment response | week 12; week 24
  the percentage of subjects achieving BASDAI50 treatment response
Change of the performance status score compared with baseline | week 12; week 24
  The performance status is used for measuring and evaluating disease activity in Ankylosing Spondylitis
Change of the spinal pain score compared with baseline | week 12; week 24
  the spinal pain is used for measuring and evaluating disease pain in Ankylosing Spondylitis
Change of morning stiffness duration compared with baseline | week 12; week 24
  The morning stiffness duration is used for measuring and evaluating disease activity in Ankylosing Spondylitis
Change of ASDAS compared with baseline | week 12; week 24
  The ASDAS is used for measuring and evaluating disease activity in Ankylosing Spondylitis
Change of BASDAI compared with baseline | week 12; week 24
  The BASDAI is used for measuring and evaluating disease activity in Ankylosing Spondylitis
Change of BASFI compared with baseline | week 12; week 24
  The BASFI consist of a set of 10 questions designed to determine the degree of functional limitation in subjects with AS. The BASFI score was derived based on the average of questions 1 through 10. The first 8 questions considered activities related to functional anatomy and the final 2 questions assessed the subject's ability to cope with everyday life over the last week. A 10 cm visual analog scale (VAS) was used to answer the questions and the mean of the ten scales gave the BASFI score a value between 0 (easy) and 10 (impossible).
Change of BASMI compared with baseline | week 12; week 24
  The BASMI measures the range of motion based on five clinical measurements: 1) cervical rotation, 2) tragus to wall distance, 3) lumbar side flexion, 4) lumbar flexion (modified Schober's) and 5) intermalleolar distance. The total BASMI score ranges from 0 to 10 reflecting mild to moderate disease activity and functional ability in the spinal column. The higher the BASMI score the more severe the patient's limitation of movement due to their ankylosing spondylitis
Change of SF-36 compared with baseline | week 12; week 24
  SF-36 survey will be used to calculate overall, mental (MCS) and physical (PCS) component scores at week 12; week 24 compared to baseline
Change of EQ-5D compared with baseline | week 12; week 24
  EQ-5D is a standard instrument to measure of health status
Change of chest expansion compared with baseline | week 12; week 24
  Chest expansion, measured in cm, is defined as the difference in thoracic circumference during full expiration versus full inspiration, measured at the fourth intercostal space (nipple line). The better of 2 tries was recorded. Higher scores indicate better health. Change from baseline greater than (>) 0 represented improvement.
Change of MASES compared with baseline | week 12; week 24
  The Maastricht Ankylosing Spondylitis Enthesitis Score quantitates inflammation of the entheses (enthesitis) by assessing pain at the following entheses (sites where tendons or ligaments insert into the bone): 1st costochondral joints left/right; 7th costochondral joints left/right; posterior superior iliac spine left/right; anterior superior iliac spine left/right; iliac crest left/right; 5th lumbar spinous process; and the proximal insertion of the Archilles tendon left/right.
Change of swollen and tender joint counts at week 12 and week 24 compared with baseline. | week 12; week 24

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No